CLINICAL TRIAL: NCT03361813
Title: Comparative Study Between Pre-emptive Trans-cutaneous Versus Trans-oral Ultrasound Guided Peritonsillar Space Infiltration With Bupivacaine During Elective Tonsillectomy
Brief Title: Pre-emptive Trans-cutaneous Versus Trans-oral Ultrasound Guided Peritonsillar Infiltration With Bupivacaine During Tonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed H Othman, Assisstant professor of Anesthesia ICU and pain Relief, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201617019.2P
Record Dates: First submitted 2017-11-19; First posted 2017-12-05 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Postoperative Pain Management

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trans-cutaneous ultrasound guided peritonsillar infiltration (Active Comparator)
  Interventions: Other: trans-oral ultrasound guided peritonsillar infiltration
- trans-oral ultrasound guided peritonsillar infiltration (Placebo Comparator)
  Interventions: Other: trans-cutaneous ultrasound guided peritonsillar infiltration

INTERVENTIONS:
Other: trans-cutaneous ultrasound guided peritonsillar infiltration — Preoperative peritonsillar infiltration of bupivacine in tonsillectomy surgery by using the ultrasound through a transcutaneous route
  Arms: trans-oral ultrasound guided peritonsillar infiltration
Other: trans-oral ultrasound guided peritonsillar infiltration — Preoperative peritonsillar infiltration of bupivacine in tonsillectomy surgery by using the ultrasound through a trans-oral route
  Arms: trans-cutaneous ultrasound guided peritonsillar infiltration

SUMMARY:
Ultrasound as a technique is safe, readily available, quick and portable allowing more accuracy of different regional blocks and local infiltration. It allows imaging of the mouth, oropharynx, infrahyoid structures, larynx, vocal cords, and trachea. Recently, ultrasound has been shown to improve accuracy in ultrasound guided block with local anesthetic infiltration. The objective of our study is to compare the effect of pre-emptive trans-oral ultrasound guided peritonsillar infiltration versus trans-cutaneous ultrasound (US) guided peritonsillar infiltration with bupivacaine for post-tonsillectomy analgesia, on surgical field, and surgeon satisfaction(intra-operative reactionary bleeding).

Materials and Methods: the patients will be admitted for tonsillectomy at ENT department of the Al- Azhar university hospitals. The patients' ages between 3 to 15 years. Patients will be divided into Cutaneous group: patients will be submitted to Trans-cutaneous ultrasound guided peritonsillar infiltration with bupivacaine, and Oral group: patients will be submitted to Trans-oral ultrasound guided peritonsillar infiltration with bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status I-II with no airway complications or systemic diseases or known psychological diseases. Reason for their surgery was recurrent or chronic tonsillitis.

Exclusion Criteria:

* Infection at the site of injection, peritonsillar abscess or cellulites.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Surgical field (intra-operative reactionary bleeding and/or muscle tear) | time of surgery
  * Iintra-operative reactionary bleeding and/or muscle tear assessment by number of soaked gauze per 20 min (per tonsil) (3 soaked gauze per 20 min (per tonsil) = no reactionary bleeding (0 point), 6 soaked gauze per 20 min (per tonsil) = mild bleeding (1 point) and 10 soaked gauze or more per 20 min (per tonsil) = moderate to severe bleeding (2 points).
  * Dissection time assessment (dissection time 10 min or less per tonsil = no bleeding (0 point), dissection time 20 min per tonsil = mild bleeding (1 point) and dissection time 30 min or more per tonsil = moderate to severe bleeding (2 points).
Surgeon satisfaction | time of surgery
  Direct surgeon questionnaire assessment about bleeding and surgical field (full satisfaction= no bleeding (0 point), fair satisfaction= mild bleeding (1point), and poor satisfaction= moderate to severe bleeding (2 points)

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University Hospital, Cairo, Egypt